CLINICAL TRIAL: NCT05191056
Title: Anti-aging and Anti-oxidant Efficacy Evaluation of the MelaGene
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TSMH IRB No. 21-057-A
Record Dates: First submitted 2022-01-04; First posted 2022-01-13 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Aging; Antioxidative Stress

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo drink (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo drink
- MelaGene drink (Experimental)
  Interventions: Dietary Supplement: MelaGene drink

INTERVENTIONS:
Dietary Supplement: Placebo drink — consume 1 bottle per day for 8 weeks
  Arms: Placebo drink
Dietary Supplement: MelaGene drink — consume 1 bottle per day for 8 weeks
  Arms: MelaGene drink

SUMMARY:
The primary purpose of the present study is to evaluate the effects of MelaGene on anti-aging and anti-oxidant.

ELIGIBILITY:
Inclusion Criteria:

* 30 to 65-year-old;
* Must read and sign the informed consent form before the experiment;
* People who are willing to cooperate with contraception during the trial period;
* Do not change lifestyle and eating habits arbitrarily during the trial period;
* Do not take supplementary foods and health supplements with the same efficacy two weeks before and during the test;
* If any adverse reaction occurs during the experiment, subjects should be notified the researcher immediately.

Exclusion Criteria:

* Subject who is not willing to participate in this study;
* Vegetarians;
* People with a history of organ transplantation, epilepsy or convulsions, liver and kidney disease, malignant tumors, endocrine diseases, mental illness, alcohol or drug abuse, and other major organic diseases (according to medical history);
* Participate in other clinical trials related to antioxidants and anti-aging four weeks before and during the test;
* People with a history of dyspepsia would affect the absorption of the test product;
* Allergic to the components of the test product;
* Pregnant or breast-feeding women;
* Take anti-oxidant supplements;
* Undergoing hormone replacement therapy.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
The change of blood lipid (Triglyceride, total cholestrol, HDL-C, LDL-C) | Days 1, 28, and 56
  Venous blood is sampled to measure concentrations of blood lipid (Triglyceride, total cholestrol, HDL-C, LDL-C)
The change of ALT and AST | Days 1, 28, and 56
  Venous blood is sampled to measure concentrations of ALT and AST
The change of MDA | Days 1, 28, and 56
  Venous blood is sampled to measure concentrations of MDA
The change of blood antioxidants(f-Thiols, t-GSH, GST-RBC, SOD, Total Anit-oxidative Capicity) | Days 1, 28, and 56
  Venous blood is sampled to measure concentrations of blood antioxidants(f-Thiols, t-GSH, GST-RBC, SOD, Total Anit-oxidative Capicity)
The change of anti-aging gene expression | Days 1, 28, and 56
  Venous blood is sampled to measure expression of anti-aging gene
The change of cardiovascular endurance | Days 1, 28, and 56
  Step test is designed to assess cardiovascular endurance

SECONDARY OUTCOMES:
The change of continuous attention test | Days 1, 28, and 56
  Continuous attention test is designed to assess cognitive performance
The change of fatigue condition | Days 1, 28, and 56
  BFI-Taiwan Form is collected to assess fatigue condition

CONTACTS AND LOCATIONS:
Overall Officials: Bo han Wu, Ph.D, Principal Investigator — Pingtung University of Science and Technology
Locations (1):
- Bo Han Wu, Pingtung City, Taiwan